CLINICAL TRIAL: NCT05372744
Title: The Influence of Expectations on Affect-regulatory Characteristics of Deceptive Placebos: An Experimental Investigation
Brief Title: Affect-regulatory Characteristics of Deceptive Placebos
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Wrief
Record Dates: First submitted 2022-05-09; First posted 2022-05-13 (Actual); Last update posted 2023-06-23 (Actual); Status verified 2023-06

CONDITIONS: Social Anxiety; Depression
MeSH Terms: conditions — Depression | interventions — Antidepressive Agents

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Experimental group (anticipatory) (Experimental): Participants receive a nasal spray that is in fact a placebo. However, they are told that it protects from experiencing intensive emotional reactions and consequent rumination tendencies. They take the nasal spray once in the laboratory.
  Interventions: Other: Active Placebo labelled as antidepressant
- Experimental group (reactive) (Experimental): Participants receive a nasal spray that is in fact a placebo. Participants of this group are told, however, that it helps to regulate experienced intensive emotional reactions and to distance oneself from consequent ruminative thoughts. They take the nasal spray once in the laboratory.
  Interventions: Other: Active Placebo labelled as antidepressant
- No-treatment control group (No Intervention): Participants do not receive the nasal spray and continue with the following task.

INTERVENTIONS:
Other: Active Placebo labelled as antidepressant — Participants receive an active nasal spray that is in fact a placebo with a specific framing in regards to its affect-regulatory characteristics, respectively.
  Arms: Experimental group (anticipatory); Experimental group (reactive)

SUMMARY:
The study tries to identify whether specifically framed expectations, induced with an active placebo nasal-spray, have effects on affective regulation processes and rumination.

DETAILED DESCRIPTION:
Healthy volunteers are informed that a new application method for an antidepressant, specialized on positively influencing the experience of aversive emotional states would be tested. They will randomly be assigned to a no treatment control group (not taking a placebo) or to one of the two treatment groups: Participants will be taking the antidepressant (which is in fact an active placebo) which will either protect them from experiencing intense emotional reactions and rumination (anticipatory group) or help them to regulate emotional states quicker as well as to distance themselves from ruminative thoughts (reactive group). Then, an aversive emotional state is induced by an autobiographical recall of events which made the participants feel inadequate, bashful, and ashamed. Currently experienced shame as well as state rumination are assessed before and after the negative recall task.

ELIGIBILITY:
Inclusion Criteria:

* healthy volunteers
* fluent in German language

Exclusion Criteria:

* mental disorders
* allergic to capsaicin
* allergic to sesame oil
* intake of psychopharmacological drugs in the last four weeks
* intake of illegal drugs in the last two weeks
* consumption of alcohol in the last twelve hours
* students in medicine, pharmacy, or psychology
* completed studies in medicine, pharmacy or psychology
* current pregnancy or lactation
* cardio vascular disease
* kidney disease
* liver disease

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 127 (Actual)
Dates: Start 2022-05-25 (Actual); Primary Completion 2022-07-31 (Actual); Study Completion 2022-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Experienced Shame (Experienced Shame Scale, 'ESS') | At baseline and after autobiographical recall. Each assessment is taking 5 minutes, in total 10 minutes.
  German questionnaire of 11 items, e.g., physical phenomena: feeling "very warm--- very cold; pale---flushed"; emotional phenomena: feeling "good---bad, clear---confused, calm---highly aroused ", social phenomena: feeling like "hiding---being sociable, talking---being quiet" All Items will be rated on a Likert scale from 1 (= strongly disagree) to 7 (= strongly agree)

SECONDARY OUTCOMES:
Change in State Rumination (Fragebogen zur Erfassung aktueller Ruminationsneigung) | At baseline and after the rumination induction. Each assessment is taking 5 Minutes, in total 10 minutes.
  German questionnaire of 10 Items, e.g.: "I get lost in ruminative thoughts.", "I am present in this situation.", "My thoughts are focused on the past.". All Items will be rated on a Likert scale from 0 (not at all) to 10 (very much).

CONTACTS AND LOCATIONS:
Locations (1):
- Philipps-Universität Marburg, Marburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Schafer LN, Rief W. The influence of expectations on shame, rumination and cognitive flexibility: an experimental investigation on affect-regulatory characteristics of deceptive placebos. Front Psychol. 2025 Jan 10;15:1502460. doi: 10.3389/fpsyg.2024.1502460. eCollection 2024. PMID 39868023